CLINICAL TRIAL: NCT07258719
Title: Aromatherapy's Impact on Test Anxiety in College Students: A Mixed Methods Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jenalee Hinds (Other)
Responsible Party: Sponsor-Investigator, Jenalee Hinds, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105250
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: Aromatherapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aromatherapy intervention 1 (Experimental): participants applying their assigned essential oil (ADAPTIV or Thinker) prior to quizzes/tests
  Interventions: Other: Essential Oil 1
- aromatherapy intervention 2 (Experimental): participants applying their assigned essential oil (ADAPTIV or Thinker) prior to quizzes/tests
  Interventions: Other: Essential Oil 2

INTERVENTIONS:
Other: Essential Oil 1 — Participants will complete short tasks before and after quizzes and tests that are part of normal coursework.
  Prior to each assessment, participants will apply aromatherapy (doTERRA ADAPTIV) using a roller bottle (Weeks 5-12 only), sit quietly for 3 minutes, and record resting Heart Rate and Blood Pressure. T After completing the quiz/test, participants will repeat HR and BP measurements and complete a brief post-assessment questionnaire.
  Other Names: ADAPTIV
  Arms: aromatherapy intervention 1
Other: Essential Oil 2 — Participants will complete short tasks before and after quizzes and tests that are part of normal coursework.
  Prior to each assessment, participants will apply aromatherapy (doTERRA Thinker) using a roller bottle (Weeks 5-12 only), sit quietly for 3 minutes, and record resting Heart Rate and Blood Pressure. T After completing the quiz/test, participants will repeat HR and BP measurements and complete a brief post-assessment questionnaire.
  Other Names: Thinker
  Arms: aromatherapy intervention 2

SUMMARY:
This study aims to investigate the effectiveness of aromatherapy as an intervention to reduce test anxiety and improve academic performance. The Investigators hypothesize that exposure to aromatherapy during assessments will lead to lower levels of test anxiety and result in higher quiz and test scores.

ELIGIBILITY:
Inclusion Criteria:

* current student
* participating in selected course at the University

Exclusion Criteria:

* allergy to essential oils
* pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-09-18 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Change in Westside Test Anxiety Scale (WTAS) | Baseline and Week 12
  The WTAS consists of 10 items, each using a Likert response scale where 1= "Never true" and 5= "always true. Total score is divided by 10 to obtain final scores. The total score ranges from one to five with higher scores equating to greater anxiety.
Change in heart rate (HR) pre aromatherapy | week 3 and week 4
  heart rate will be measured with a fitness tracker before and after quizzes/tests
Change in blood pressure (BP) pre aromatherapy | week 3 and week 4
  both systolic and diastolic blood pressure will be measured with a fitness tracker before and after quizzes/tests
Change in heart rate (HR) with aromatherapy | Week 5 through Week 12
  heart rate will be measured with a fitness tracker before and after quizzes/tests
Change in blood pressure (BP) with aromatherapy | Week 5 through Week 12
  both systolic and diastolic blood pressure will be measured with a fitness tracker before and after quizzes/tests
Change in Stress Performance Evaluation (SPE) | Baseline and week 12
  percent test questions correct (number of test questions correct out of hundred)]/ percent change in heart rate (heart rate at baseline)/(heart rate after testing) × 100)]

CONTACTS AND LOCATIONS:
Overall Officials: Jenalee Hinds, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No